CLINICAL TRIAL: NCT06959758
Title: Effects of Probiotics (BioKid LR - Contains Nine Different Species of Probiotics Bacteria Including L. Reuteri) in Children With Functional Constipation: a Double Blind Randomized Control Trial
Brief Title: Effects of Probiotics (BioKid LR - Contains Nine Different Species of Probiotics Bacteria Including L. Reuteri) in Children With Functional Constipation
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ferass Abu Hanna (Other)
Collaborators: Ambrosia - SupHerb Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Ferass Abu Hanna, Principal Investigator, HaEmek Medical Center, Israel
Organization: HaEmek Medical Center, Israel (Other)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 0151-23-EMC
Record Dates: First submitted 2025-05-05; First posted 2025-05-07 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-04

CONDITIONS: Constipation
Keywords: constipation; laxatives; PEG 350
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BioKid Arm (Experimental): This arm includes children receiving the BioKid LR probiotic supplement alongside standard laxative treatment (PEG 3350), followed by BioKid LR alone after PEG tapering.
  Interventions: Dietary Supplement: Probiotic Arm
- Placebo (Placebo Comparator): This arm includes children receiving a placebo (maltodextrin powder) alongside standard laxative treatment (PEG 3350), followed by placebo alone after PEG tapering.
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic Arm — It is administered daily to children with functional constipation, alongside standard laxative treatment (PEG 3350) for the first 12 weeks, and then continued alone for the remainder of the 52-week study period. The study evaluates whether BioKid LR® helps maintain normal bowel movements after stopping PEG.
  Arms: BioKid Arm
Drug: Placebo — A placebo maltodextrin powder is administered daily to children with functional constipation, alongside standard laxative treatment (PEG 3350) for the first 12 weeks, and then continued alone for the remainder of the 52-week study period.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate whether a probiotic supplement, BioKid LR®, can help maintain normal bowel movements after stopping laxative treatment (PEG 3350) in children aged 6 months to 17 years with functional constipation.

The main questions it aims to answer are:

Does taking BioKid LR reduce the chance of constipation coming back after stopping PEG? Can BioKid LR help children maintain regular bowel movements without needing to restart laxatives? Researchers will compare children who take BioKid LR with those who take a placebo (an inactive powder) to see if the probiotic helps prevent constipation from returning.

Participants will:

Take PEG 3350 (a common laxative) for 12 weeks along with either BioKid LR or a placebo.

After 12 weeks, begin gradually stopping PEG while continuing with BioKid LR or placebo for another 12 weeks.

Then continue only with BioKid LR or placebo for an additional 28 weeks (total study duration: 52 weeks).

Keep a stool diary to track bowel habits and any side effects. Attend 5 study visits for physical exams and monitoring (weeks 0, 12, 24, 38, 52).

The study includes 80 children and is double-blinded, meaning neither the doctors nor the participants know who is receiving the real probiotic or the placebo.

The primary outcome is how long it takes for constipation to return after stopping PEG, requiring retreatment.

Secondary outcomes include:

How many children still need long-term treatment. How many have regular bowel movements without accidents (in children over 4 years old).

Stool consistency and frequency. Children with certain medical conditions (like celiac disease or hypothyroidism) or who are taking medications that cause constipation cannot participate.

This study is supported by Supherb Group, Israel, but they are not involved in designing or analyzing the research. The study has been approved by an ethics committee and follows international ethical guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Age 0.5 - 17 years
2. Diagnosis of FC based on Rome IV criteria

Exclusion Criteria:

1. Children with chronic diseases which could cause constipation: Celiac disease, food allergy, Hypothyroidism, Inflammatory Bowel Disease, electrolytes disturbances, Cystic fibrosis, Hirschsprung disease, Neuropathic conditions (Spinal cord trauma, Neurofibromatosis, Tethered cord) or intestinal pseudo-obstruction
2. Prematurity (<34 weeks)
3. S/P intestinal surgery
4. Immunodeficiency
5. Malignancy
6. Children treated with medications associated with constipation. *

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Constipation Recurrence | 52 weeks
  Time to recurrence of constipation after PEG withdrawal necessitating retreatment with PEG.
  This measures how long it takes for constipation to return after stopping laxative treatment, requiring the child to start PEG again.

SECONDARY OUTCOMES:
Intractable Constipation | 12 weeks
  Prevalence of intractable constipation after the initial 12 weeks of PEG treatment
Normal Bowel Movements without PEG | 52 weeks
  Failure to maintain normal bowel movements (defined as > 3 spontaneous bowel movement per week) with no fecal incontinence (among children older than 4 year old) without necessitating PEG re-treatment, at weeks 24 and 52.

CONTACTS AND LOCATIONS:
Locations (1):
- Emek Medical Center, Afula, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Eskesen D, Jespersen L, Michelsen B, Whorwell PJ, Muller-Lissner S, Morberg CM. Effect of the probiotic strain Bifidobacterium animalis subsp. lactis, BB-12(R), on defecation frequency in healthy subjects with low defecation frequency and abdominal discomfort: a randomised, double-blind, placebo-controlled, parallel-group trial. Br J Nutr. 2015 Nov 28;114(10):1638-46. doi: 10.1017/S0007114515003347. Epub 2015 Sep 18. PMID 26382580
- [Background] Banaszkiewicz A, Szajewska H. Ineffectiveness of Lactobacillus GG as an adjunct to lactulose for the treatment of constipation in children: a double-blind, placebo-controlled randomized trial. J Pediatr. 2005 Mar;146(3):364-9. doi: 10.1016/j.jpeds.2004.10.022. PMID 15756221
- [Background] Modin L, Walsted AM, Rittig CS, Hansen AV, Jakobsen MS. Follow-up in Childhood Functional Constipation: A Randomized, Controlled Clinical Trial. J Pediatr Gastroenterol Nutr. 2016 Apr;62(4):594-9. doi: 10.1097/MPG.0000000000000974. PMID 26348685
- [Background] Bongers ME, van Wijk MP, Reitsma JB, Benninga MA. Long-term prognosis for childhood constipation: clinical outcomes in adulthood. Pediatrics. 2010 Jul;126(1):e156-62. doi: 10.1542/peds.2009-1009. Epub 2010 Jun 7. PMID 20530072
- [Background] Tabbers MM, DiLorenzo C, Berger MY, Faure C, Langendam MW, Nurko S, Staiano A, Vandenplas Y, Benninga MA; European Society for Pediatric Gastroenterology, Hepatology, and Nutrition; North American Society for Pediatric Gastroenterology. Evaluation and treatment of functional constipation in infants and children: evidence-based recommendations from ESPGHAN and NASPGHAN. J Pediatr Gastroenterol Nutr. 2014 Feb;58(2):258-74. doi: 10.1097/MPG.0000000000000266. PMID 24345831
- [Background] Mugie SM, Benninga MA, Di Lorenzo C. Epidemiology of constipation in children and adults: a systematic review. Best Pract Res Clin Gastroenterol. 2011 Feb;25(1):3-18. doi: 10.1016/j.bpg.2010.12.010. PMID 21382575